CLINICAL TRIAL: NCT00802386
Title: Screening for Bacterial Vaginosis Screening at IUD Insertion: Is There a Role?
Brief Title: Bacterial Vaginosis Screening at IUD Insertion
Status: Completed | Type: Observational
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 07-358
Record Dates: First submitted 2008-12-03; First posted 2008-12-04 (Estimated); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: BACTERIAL VAGINOSIS
Keywords: BACTERIAL VAGINOSIS; IUD INSERTION
MeSH Terms: conditions — Vaginosis, Bacterial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — WHOLE BLOOD; VAGINAL SWAB
Oversight: Data Monitoring Committee: No

SUMMARY:
A number of studies have shown a higher prevalence of BV among IUD users.13,,14 None, however, have screened women prior to inserting the IUD. No data exists detailing the status of the vaginal microflora and possible cervical infection prior to IUD insertion. Thus, no inference can be made about the possible influence of IUD insertion and presence to the development of upper genital tract infection . Consequently, with the current literature, it would be difficult to make an argument for screening and treatment for BV prior to IUD insertion. This study will help us determine whether women with an IUD develop a change in the normal bacteria that are present in the vagina, known as bacterial vaginosis (BV). In addition, in those women with BV, we are looking to see if they develop more significant problems with the IUD, than those who do not have BV. Overall, this will help us determine whether all women should be screened for BV prior to IUD insertion.

ELIGIBILITY:
Inclusion Criteria:

* Women between the ages of 18 and 48, who request to have an IUD inserted, both for contraceptive and noncontraceptive indications, will be asked to participate in the study.

Exclusion Criteria:

* pregnancy
* a previous history of ectopic pregnancy or pelvic inflammatory disease
* HIV positive or immunocompromised
* unable to understand English
* unable to give informed consent

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women between the ages of 18 and 48, who request to have an IUD inserted, both for contraceptive and noncontraceptive indications, will be asked to participate in the study.
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2008-01; Primary Completion 2009-03 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Rate of abnormal bleeding | 1 month
  In the study population, we will calculate the number of women who have BV at the time of IUD insertion. In order to assess abnormal bleeding, participants will be asked to keep a menstrual calendar denoting the bleeding characteristics (heavy, normal, light flow or spotting).
Pain/cramping | 1 month
  Participants will be asked to monitor for any signs or symptoms of infection, such as pelvic pain, foul purulent discharge or fever > 38oC.
Expulsion | 1 month
  At the 1-month follow-up visit, repeat swabs for BV will be taken and we will also checking that the IUD is still in place, by the presence of visible IUD strings at the cervical os.
Pelvic infection | 1 month
  Participants will be asked to monitor for any signs or symptoms of infection, such as pelvic pain, foul purulent discharge or fever > 38oC.

SECONDARY OUTCOMES:
Occurence of new onset BV infection | 1 month post-IUD insertion
  We will look at women who did not have BV at the first visit but who acquire this infection at the 1-month visit. From this, we may make an inference about the possible influence of IUD insertion and presence on the occurrence of vaginal flora changes.

CONTACTS AND LOCATIONS:
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada